CLINICAL TRIAL: NCT06846151
Title: Clinical Investigation of Optos OCT in Patients with Retinal Pathologies
Brief Title: Retinal Investigation Using Optos OCT Device
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Optos, PLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OPT1105; REC ref: 25/NS/0018 (Other: The North of Scotland Research Ethics Committee); IRAS Project ID: 338297 (Other: Integrated Research Application System)
Record Dates: First submitted 2025-02-13; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: AMD - Age-Related Macular Degeneration; Retinitis Pigmentosa (RP); Diabetic Retinopathy; Control Patients
MeSH Terms: conditions — Macular Degeneration; Retinitis Pigmentosa; Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: all participants receive a single intervention at a single point in time
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- standard imaging process (Other): All participants will undergo the same imaging
  Interventions: Device: retinal functional imaging

INTERVENTIONS:
Device: retinal functional imaging — this is a proof of concept study
  Other Names: OCT

SUMMARY:
Retinal investigation using OCT with control and diseased eyes

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants 18 years of age or older who have full legal capacity to volunteer on the date the informed consent is signed.
2. Participants who understand the study and patient information sheet and can follow the instructions.
3. Participants who agree to participate in the study.
4. Control group where no retinal abnormalities were detected as part of the standard basic ophthalmic examination.
5. Participants with retinal disease in at least one eye including: Early dry age-related macular degeneration, late stage dry age-related macular degeneration specifically geographic atrophy, Wet age-related macular degeneration, Retinitis pigmentosa, Diabetic retinopathy and other macular atrophic diseases

Exclusion Criteria:

1. Inability to understand written and verbal English sufficiently to comprehend the study and provide informed consent
2. Ophthalmic disease other than condition under investigation.
3. Participants unable to tolerate ophthalmic imaging.
4. Cataract (unless deemed mild in the opinion of the investigator)
5. Participants with significant ocular media not sufficiently clear to obtain acceptable OCT images.
6. Diabetes (unless part of the diabetic eye disease group)
7. Binocular visual acuity worse than 6/18
8. Strabismus (squint)
9. Age related macular degeneration groups: polypoidal choroidal vasculopathy
10. Participants with photo sensitivity epilepsy, experience of seizures, or sensitivity to flickering light (based on self-report)
11. Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
OCT physical response data | 6 months from recruitment start
  Response data per participant will be collected and analyzed